CLINICAL TRIAL: NCT02936960
Title: Endoscopic Ultrasound-guided Needle-based Confocal Laser Endomicroscopy in Solid Pancreatic Masses
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2016SDU-QILU-20
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Solid Pancreatic Masses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The differential diagnosis of solid pancreatic masses by endoscopic ultrasound-guided fine-needle aspiration (EUS-FNA) is currently suboptimal. Needle-based confocal laser endomicroscopy (nCLE) is a novel endoscopic technique, which is compatible with the 19-gauge FNA needle. Under endoscopic ultrasonography (EUS) guidance, nCLE enables real-time in vivo imaging of lesion tissues at cellular and subcellular levels. This study aimed to describe nCLE interpretation criteria for the characterization of pancreatic masses, with histopathological correlation, and to perform the validation of these criteria.

ELIGIBILITY:
Inclusion Criteria:

* patients with any pancreatic mass

Exclusion Criteria:

* Patients aged <18 years or >80 years
* Known allergy to fluorescein dye
* Previous EUS-FNA performed within the past 3 months, and usualcontraindications to EUS-FNA
* Pregnancy or breastfeeding
* Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients undergoing EUS for the diagnosis and staging of a pancreatic mass will be recruited in this study at Qilu Hospital, Shandong University.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The nCLE interpretation criteria for the characterization of pancreatic masses with histopathological correlation | 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD. MD., Study Director — Department of Gastroenterology, Qilu Hospital, Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China